CLINICAL TRIAL: NCT02535806
Title: A Pilot Study of Mitoxantrone-Based Four Drug Reinduction in Combination With Bortezomib for Relapsed or Refractory Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma in Children and Young Adults
Brief Title: Four Drug Reinduction With Bortezomib for Relapsed or Refractory ALL or LL in Children and Young Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding source discontinued
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Keith August, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MERCY01
Record Dates: First submitted 2015-08-04; First posted 2015-08-31 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: Relapsed, Refractory
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Bortezomib; Methotrexate; Hydrocortisone; Cytarabine; Dexamethasone; Mitoxantrone; Vincristine; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Treatment Arm (Experimental): Velcade will be given IV push on days 1,4,8 and 11 at a dose of 1.3 mg/m2/dose. At least 72 hours must have relapsed between doses.
  IT Methotrexate (CNS Negative patients only) on days 1 and 8; age based dosing IT Methotrexate/Hydrocortisone/AraC (CNS positive patients only) on days 1, 8, 15 and 22; age based dosing.
  Dexamethasone: Days 1-5 and 15-19; 10mg/m2/dose PO BID. Mitoxantrone: Days 1 and 2; 10mg/m2/dose Vincristine: days 1, 8, 15, and 22 at 1.5 mg/m2 (Maximum dose 2 mg) PEG-asparaginase: Days 3 and 17, 2500 IU/m2/dose
  Interventions: Drug: Velcade; Drug: Methotrexate; Drug: Methotrexate / Hydrocortisone / Cytarabine; Drug: Dexamethasone; Drug: Mitoxantrone; Drug: Vincristine; Drug: Pegaspargase

INTERVENTIONS:
Drug: Velcade — 4 doses of study drug will be given.
  Other Names: Bortezomib
Drug: Methotrexate — Intrathecal dose For CNS negative patients, Day 1 and Day 8
Drug: Methotrexate / Hydrocortisone / Cytarabine — Intrathecal dose for CNS positive patients, Day 1, 8, 15, 22
Drug: Dexamethasone — Days 1-5 and 15-19
Drug: Mitoxantrone — Days 1 and 2
Drug: Vincristine — Days 1, 8, 15, 22
Drug: Pegaspargase — Days 3 and 17

SUMMARY:
This is a phase II study designed to investigate the combination of bortezomib with the mitoxantrone reinduction regimen used in the ALL R3 trial. The study will enroll patients with high risk ALL relapse including early bone marrow relapse and second or greater relapse of any kind. Patients with relapsed LL will also be eligible. Bone marrow evaluation will be performed after blood counts recover to assess the rate of CR (<5% bone marrow blasts) and MRD status in children following this regimen. Further treatment with or without HSCT will be at the discretion of the primary physician.

DETAILED DESCRIPTION:
1.0 GOALS AND OBJECTIVES (SCIENTIFIC AIMS)

1.1 Primary Aims

1.1.1 To evaluate the feasibility and toxicity of using bortezomib in combination with the ALL R3 re-induction regimen in pediatric patients with relapsed or refractory ALL or LL.

1.1.2 To determine the rate of complete response and negative minimal residual disease status following bortezomib combined with R3 reinduction.

2.0 BACKGROUND

Despite the progress that has been made in the treatment of ALL in children, relapse of disease remains a significant treatment problem. By itself, the number of patients with relapsed ALL would be the 4th most common childhood malignancy and overall survival in these patients is poor. Using conventional treatments, second remission rates after bone marrow relapse in ALL are 81-93% and long-term event free survival (EFS) is only 27-50%. Initial standard therapy for children following relapse includes a four drug reinduction strategy, typically using prednisone, vincristine, PEG-asparaginase, and doxorubicin. For children with first marrow relapse of ALL less than 36 months from diagnosis, this four drug reinduction strategy results in a CR rate of 68%. However, 75% of patients in CR2 had minimal residual disease (MRD) that was positive (>0.01%) at the end of reinduction. The presence of MRD in relapsed ALL is strongly associated with worse long term outcomes. For children with ALL that relapsed following a second (CR2) remission, outcomes are dismal with 5 year disease free survival of 15%.

In 2010, results were published of the ALL R3 trial from the Children's Cancer and Leukemia Group in the United Kingdom and Ireland. This trial randomized children with first relapse of ALL to receive a four drug reinduction using either mitoxantrone or idarubicin as the anthracycline. The study was closed early due to a statistically significant improvement in survival for children randomized to mitoxantrone. Children who received mitoxantrone had a 3 year disease free survival of 64.6% compared to 35.9% in the idarubicin group. Toxicities in this study were not excessive, and children randomized to receive mitoxantrone had significantly less toxicity than those in the idarubicin group. Based on the results of this trial, the Children's Oncology Group (COG) has begun using this reinduction regimen as the backbone for new clinical trials for children with relapsed ALL.

Despite the improvement in outcomes for the children with relapsed ALL treated with mitoxantrone on the R3 study, there is still a need for continued efforts to improve outcomes in patients with ALL and LL that experience a relapse. This is particularly true for high risk groups such as those who have an early bone marrow relapse (<36 months from diagnosis), second or greater relapse or relapsed LL where long term survival remains less than 50% Bortezomib is a proteasome inhibitor that has demonstrated activity in a number of cancer types including acute leukemias. Bortezomib acts by inhibiting the ubiquitin-proteasome pathway resulting in the blockade of NF-κB activation and the stabilization of multiple proapoptotic proteins including p53, p21, p27, and Bax. Collectively, these effects induce apoptosis and enhance the cytotoxic effects of chemotherapy. In the Pediatric Preclinical Testing Program (PPTP), bortezomib showed activity against a number of ALL cell lines. As a single agent, bortezomib was effective at inhibiting NF-κB but there was no clinical response in 9 heavily pretreated children with ALL. Proteasome inhibition is able to induce apoptosis, and may be best utilized in combination with other conventional chemotherapy drugs to help overcome resistance. Preclinical evaluation of bortezomib with a number of drugs commonly used in pediatric ALL therapy demonstrated synergy with dexamethasone and additive effects when given along with vincristine, asparaginase, and doxorubicin.

In a phase 1 study of children with relapsed ALL of bortezomib combined with a four drug reinduction using dexamethasone, vincristine, doxorubicin, PEG-asparaginase and intrathecal therapy, bortezomib at a dose of 1.3 mg/m2 given on days 1, 4, 8 and 11 was well tolerated. The phase 2 study of this regimen was able to produce a complete response or complete response without platelet recovery in 73% of patients. These results are encouraging as these were heavily pretreated patients treated with 2 or 3 previous regimens. Due to 3 deaths from infectious toxicities, the study was amended to require infectious prophylaxis with vancomycin, levofloxacin, and voriconazole. No further deaths were seen in children following this change. Other toxicities seen on this study include grade 3 peripheral neuropathy in 2 patients.

This is a phase II study designed to investigate the combination of bortezomib with the mitoxantrone reinduction regimen used in the ALL R3 trial. The study will enroll patients with high risk ALL relapse including early bone marrow relapse and second or greater relapse of any kind. Patients with relapsed LL will also be eligible. Bone marrow evaluation will be performed after blood counts recover to assess the rate of CR (<5% bone marrow blasts) and MRD status in children following this regimen. Further treatment with or without HSCT will be at the discretion of the primary physician.

2.1 Bortezomib for Injection 2.1.1 Scientific Background Bortezomib for Injection is a small-molecule proteasome inhibitor developed by Millennium Pharmaceuticals, Inc., (Millennium) as a novel agent to treat human malignancies. Bortezomib is currently approved by the United States Food and Drug Administration (US FDA) for the treatment of patients with multiple myeloma (MM). It is also indicated for the treatment of patients with mantle cell lymphoma (MCL) who have received at least 1 prior therapy. In the European Union (EU), bortezomib in combination with melphalan and prednisone is indicated for the treatment of patients with previously untreated MM who are not eligible for high-dose chemotherapy with bone marrow transplant. Bortezomib is indicated as monotherapy for the treatment of progressive MM in patients who have received at least 1 prior therapy and who have already undergone or are unsuitable for bone marrow transplantation.

By inhibiting a single molecular target, the proteasome, bortezomib affects multiple signaling pathways. The antineoplastic effect of bortezomib likely involves several distinct mechanisms, including inhibition of cell growth and survival pathways, induction of apoptosis, and inhibition of expression of genes that control cellular adhesion, migration, and angiogenesis. Thus, the mechanisms by which bortezomib elicits its antitumor activity may vary among tumor types, and the extent to which each affected pathway is critical to the inhibition of tumor growth could also differ. Bortezomib has a novel pattern of cytotoxicity in National Cancer Institute (NCI) in vitro and in vivo assays.(19) In addition, bortezomib has cytotoxic activity in a variety of xenograft tumor models, both as a single agent and in combination with chemotherapy and radiation. Notably, bortezomib induces apoptosis in cells that over express bcl-2, a genetic trait that confers unregulated growth and resistance to conventional chemotherapeutics.

The mechanisms of action leading up to apoptosis have been more clearly defined and include initiation of the unfolded protein response and direct/indirect effects on various molecular targets including cell cycle control proteins p27 and p21, cyclins, signal transduction molecules, transcription factors c-jun and HIF1-, tumor suppressor protein p53, angiogenesis factors, and many others. Bortezomib is thought to be efficacious in multiple myeloma via its inhibition of nuclear factor B (NF-B) activation, its attenuation of interleukin-6 (IL-6)-mediated cell growth, a direct apoptotic effect, and possibly anti-angiogenic and other effects.

ELIGIBILITY:
Inclusion Eligibility Criteria

* Age: > 1 and < 40 years of age at the time of enrollment
* Diagnosis: Precursor B-cell ALL with bone marrow (BM) or combined BM/extramedullary relapse; T-cell ALL with relapsed disease; LL with relapsed disease, or ALL(T or pre-B) with primary refractory disease after at least two regimens
* Performance Score: 50% for patients
* Prior Therapy Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study.

Patients who relapse on therapy other than standard ALL maintenance therapy must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. In addition, the following requirements must be met:

Cytotoxic therapy: At least 14 days since the completion of cytotoxic therapy with the exception of hydroxyurea, which is permitted up to 24 hours prior to the start of protocol therapy.

Biologic (anti-neoplastic) agent: At least 7 days since the completion of therapy with a biologic agent or donor lymphocyte infusions (DLI).

Stem cell transplant or rescue: No evidence of active graft-vs-host disease (GVHD) and ≥ 4 months must have elapsed from time of transplant. Must not be receiving GVHD prophylaxis.

* Adequate Organ Function Requirements
* Reproductive Function: Female patients of childbearing potential must have a negative pregnancy test confirmed within 2 weeks prior to enrollment, must agree not to breastfeed their infants while on this study.Male and female patients of child-bearing potential must agree to use 2 effective methods of contraception approved by the investigator, at the same time, from the time of signing the informed consent form and for a minimum of 6 months after study treatment, or agree to completely abstain from heterosexual intercourse.
* Signed written informed consent. Assent from children will be obtained per institutional guidance.

Exclusion Eligibility Criteria

* known allergy to any of the drugs on the study with the exception of PEG-asparaginase
* Isolated CNS or isolated testicular disease
* Systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The patient needs to be off pressors and have negative blood cultures for 48 hours.
* Known optic nerve and/or retinal involvement
* Patients with concomitant genetic syndrome
* Cumulative prior anthracycline exposure must not exceed 400 mg/m2
* Patients who have previously received bortezomib or other proteasome inhibitors
* Patients taking anticonvulsants known to activate the cytochrome p450 system
* Patients who cannot receive any asparaginase products
* Patients who are pregnant or breast-feeding
* Patients with planned non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* Significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with the protocol treatment or procedures, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients with myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Diagnosed or treated for another malignancy within 2 years of enrollment
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.Radiation therapy within 3 weeks before randomization.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith J August, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
We hope to publish results

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Velcade will be given IV push on days 1,4,8 and 11 at a dose of 1.3 mg/m2/dose. At least 72 hours must have relapsed between doses.
  IT Methotrexate (CNS Negative patients only) on days 1 and 8; age based dosing IT Methotrexate/Hydrocortisone/AraC (CNS positive patients only) on days 1, 8, 15 and 22; age based dosing.
  Dexamethasone: Days 1-5 and 15-19; 10mg/m2/dose PO BID. Mitoxantrone: Days 1 and 2; 10mg/m2/dose Vincristine: days 1, 8, 15, and 22 at 1.5 mg/m2 (Maximum dose 2 mg) PEG-asparaginase: Days 3 and 17, 2500 IU/m2/dose
  Velcade: 4 doses of study drug will be given.
  Methotrexate: Intrathecal dose For CNS negative patients, Day 1 and Day 8
  Methotrexate / Hydrocortisone / Cytarabine: Intrathecal dose for CNS positive patients, Day 1, 8, 15, 22
  Dexamethasone: Days 1-5 and 15-19
  Mitoxantrone: Days 1 and 2
  Vincristine: Days 1, 8, 15, 22
  Pegaspargase: Days 3 and 17
Period: Overall Study
Arm/Group | Treatment Arm
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 8 [4 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subject With Adverse Events
Description: Toxicities were assessed and graded according to CTCAE v 4.0.
Time Frame: 36 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Remission Rate Seen With Using Bortezomib in Combination With the ALL R3 Re-induction Regimen in Pediatric Patients With Relapsed or Refractory ALL or LL.
Description: Number of patients with bone marrow blast percentage <5% after treatment
Time Frame: 36 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Post-induction Level of Minimal Residual Disease Seen With Using Bortezomib in Combination With the ALL R3 Re-induction Regimen in Pediatric Patients With Relapsed or Refractory ALL or LL.
Description: Percent of Cells Positive for Minimal residual disease measured by multiparameter flow cytometry
Time Frame: 36 days
Measure: Mean (Full Range); unit: Percentage of Cells Positive for MRD
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Percentage of Cells Positive for MRD | 0.65 [0 to 1.3]

4. Secondary Outcome: 2-year Overall Survival Seen With Using Bortezomib in Combination With the ALL R3 Re-induction Regimen in Pediatric Patients With Relapsed or Refractory ALL or LL.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: 36 days
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02535806/Prot_SAP_000.pdf